CLINICAL TRIAL: NCT02484989
Title: UK Surveillance of Treated Retinopathy of Prematurity
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DALA1012
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retinopathy of prematurity: Any baby with ROP who is treated or referred to another unit for treatment either in the form of laser therapy, cryotherapy, antiVEGF agent or vitrectomy/scleral buckling (or a combination of above treatments)
  Interventions: Other: Surviellance card

INTERVENTIONS:
Other: Surviellance card

SUMMARY:
Currently, there is little recent data on regional variations in treatment methods, neonatal units that provide retinopathy (ROP) treatment, facilities for treatment available at each unit including anaesthetic support for such preterm babies, facilities to transfer babies to units that offer treatment etc. While some parts of the UK have established neonatal networks and agreements among units for ROP treatment, in other parts, such arrangements are illdefined.

The number of babies needing ROP treatment may be higher since the introduction of revised guidelines in 2008 as earlier treatment has been shown to be beneficial. Collecting epidemiological data through the British Ophthalmic Surveillance Unit (BOSU) on the incidence of treatable ROP, the treatment methods used and facilities for treatment will provide the foundation for effective planning of resources and manpower to deal with the additional demand.

ELIGIBILITY:
Inclusion Criteria:

* Any baby with ROP who is treated or referred to another unit for treatment either in the form of laser therapy, cryotherapy, antiVEGF agent or vitrectomy/scleral buckling (or a combination of above treatments)

Exclusion Criteria:

* None; we will monitor data to exclude duplication of cases which may arise from children being transferred between neonatal units or consultants

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies with retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of babies requiring treatment for retinopathy of prematurity in the UK | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Dahlmann-Noor, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, London, United Kingdom

REFERENCES:
- [Derived] Adams GG, Bunce C, Xing W, Butler L, Long V, Reddy A, Dahlmann-Noor AH. Treatment trends for retinopathy of prematurity in the UK: active surveillance study of infants at risk. BMJ Open. 2017 Mar 21;7(3):e013366. doi: 10.1136/bmjopen-2016-013366. PMID 28325857